CLINICAL TRIAL: NCT03600831
Title: A Randomized Phase Ⅱ/Ⅲ Trial of Postoperative Concurrent Chemoradiotherapy Versus Radiotherapy Alone for Patients With Locoregionally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Postoperative Concurrent Chemoradiotherapy Versus Radiotherapy Alone for Patients With Locoregionally Advanced Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Huai'an First People's Hospital (Other)
Collaborators: The Second People's Hospital of Huai'an (Other); lian shui county People's Hospital (Unknown); xuyi People's Hospital (Unknown); Chinese People's Liberation Army No. 82 Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: huaianzhuweiguo
Record Dates: First submitted 2018-07-03; First posted 2018-07-26 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal neoplasma; adjuvant therapy; chemotherapy; radiotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Docetaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- concurrent chemoradiotherapy group (Experimental): All patients in this group will receive concurrent chemoradiotherapy with DP regimen (docetaxel plus cisplatin).
  Interventions: Drug: Docetaxel plus cisplatin; Radiation: radiotherapy
- radiotherapy group (Active Comparator): All patients in this group will receive radiotherapy alone 50Gy (2.0 Gy/fraction, 5 days a week).
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Drug: Docetaxel plus cisplatin — cisplatin 25mg/m2 on day 1 and docetaxel 25mg/m2 on day 1 weekly for 5 weeks
  Arms: concurrent chemoradiotherapy group
Radiation: radiotherapy — radiotherapy: 50Gy (2.0 Gy/fraction, 5 days a week)

SUMMARY:
The aim of this study is to investigate the effect of postoperative concurrent chemoradiotherapy versus radiotherapy alone for patients with locally advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. biopsy-confirmed esophageal squamous cell carcinoma
2. age ≤ 70 years old,
3. Karnofsky performance status ≥ 70,
4. R0 esophagectomy according to the pathological examination of the resected specimens,
5. postoperative stage Ⅱ-Ⅳa according to the AJCC 7th edition of tumor-node-metastasis (TNM) classification for esophageal carcinoma
6. Adequate organ functions (1).white blood cell (WBC) ≥3×109⁄L; (2).Absolute neutrophil counts (ANC) ≥1.5×109⁄L; (3).Hemoglobin (Hb) ≥10g⁄dl; (4).Platelet (Plt) ≥100×109⁄L; (5).Total bilirubin <1.5 upper limit of normal (ULN); (6).Aspartate transaminase (AST) ≤2.5 ULN; (7).Alanine aminotransferase (ALT) ≤2.5 ULN; (8).Creatinine ≤1.5 ULN; (9).adequate pulmonary function (FEV1>0.8 L;.
7. no previous treatment or severe complications
8. Written informed consent

Exclusion Criteria:

1. previous treatment with chemotherapy or radiotherapy
2. greater than 3 months after surgery
3. complete esophageal obstruction after surgery, esophageal perforation;
4. other malignant tumors, except for skin basal cell carcinoma, or cervical carcinoma in situ, who survived with no evidence disease for over 3 years;
5. pregnant or breast-feeding women；
6. patients with any serious concurrent disease, such as severe diabetes, uncontrolled hypertension, serious chronic obstructive pulmonary disease；
7. drug addiction, Alcoholism or AIDS;
8. uncontrolled seizures or psychiatric diseases, loss of control over their own behavior;
9. with clear chemotherapy drug allergy
10. participation in other interventional clinical trials within 30 days;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | From date of randomization to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  From the date of randomization to the date of first observation of disease progression, or relapse, or death due to any cause。

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization to death from any cause, assessed up to 3 years
  From the date of randomization until the date of death
treatment-related toxicities | From the date of randomization until six months after treatment completion
  Toxicities were graded according to the National Cancer Institute Common Toxicity Criteria (NCICTC), version 3.0
Quality of life(QOL) | 1 year
  Quality of life of patient will be evaluated using EORTC QLQ-C30. Evaluation of quality of life will be performed every 3 months.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Chinese Peiple's Liberation Army No.82 Hospital, Huai'an, Jiangsu
  - Huai'an second peiple's Hospital, Huai'an, Jiangsu
  - Lianshui County Peoples Hospital, Huai'an, Jiangsu
  - xuyi peiple's Hospital, Xucheng, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided